CLINICAL TRIAL: NCT00530751
Title: Patient Perspectives on Sharing Family Medical Histories
Brief Title: Views on Sharing Family Medical History in Healthy Women Undergoing Mammograms or Breast Evaluation
Status: Withdrawn | Type: Observational
Why Stopped: PI left
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Christian Simon, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE1Z07; P30CA043703 (NIH); CASE1Z07 (Other: Case Comprehensive Cancer Center); CASE-1Z07-CC220
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention — Participants undergo a 45-60 minute interview to assess their attitudes and concerns about providing family medical history online for genetic risk assessment or research. Participants' feelings about whether or not to use an online genetic assessment tool (i.e., Genetic Risk Easy Assessment Tool [GREAT]) are explored.

SUMMARY:
RATIONALE: Learning about the concerns that individuals may have about providing family medical history online for genetic risk assessment or research may help doctors plan future research.

PURPOSE: This clinical trial is studying views on sharing family medical history in healthy women undergoing mammograms or breast evaluation.

DETAILED DESCRIPTION:
OBJECTIVES:

* To gain an initial understanding of the ethical, family, and related concerns that individuals may have when offered the option of providing family medical history online for genetic risk assessment or research.
* To identify specific directions for future research into the ethics of online genetic risk assessment.

OUTLINE: Participants undergo a 45-60 minute interview to assess their attitudes and concerns about providing family medical history online for genetic risk assessment or research. Participants' feelings about whether or not to use an online genetic assessment tool (i.e., Genetic Risk Easy Assessment Tool [GREAT]) are explored. The GREAT allows for the electronic creation, analysis, and dissemination of family histories of individuals who may be at risk for various types of cancer. Key factors influencing a participant's use of the tool, including concerns about confidentiality, privacy, informed consent, access to risk information, and security of online family history databases, are explored. Ethical issues regarding communication and agreement among family members on disclosing family medical history are also discussed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy women undergoing mammograms or being evaluated for a breast concern at the University Hospitals Breast Center

PATIENT CHARACTERISTICS:

* Able to speak English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Participants' perspectives and concerns regarding online genetic risk assessment or research
Identification of directions for future research into the ethics of online genetic risk assessment or research

CONTACTS AND LOCATIONS:
Overall Officials: Christian Simon, PhD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (7):
- United States (7):
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Geauga Regional Hospital, Chardonr, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange Villager, Ohio
  - University Suburban Health Center, South Euclid, Ohio
  - UHHS Westlake Medical Center, Westlaker, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00530751?term=NCT00530751&rank=1